CLINICAL TRIAL: NCT01269190
Title: Wide-Field and High Resolution In Vivo Imaging of Oral Neoplasia Using Topical Fluorescent Dyes: A Feasibility Study
Brief Title: Wide-Field and High Resolution In Vivo Imaging in Visualizing Lesions in Patients With Oral Neoplasia Undergoing Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008-0613; NCI-2015-01904 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2008-0613 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2010-12-30; First posted 2011-01-04 (Estimated); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Oral Cavity Neoplasm
MeSH Terms: conditions — Mouth Neoplasms | interventions — Proflavine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (widefield multispectral imaging and HRME) (Experimental): Patients undergo evaluation of oral cavity using a widefield multispectral imaging device and a high-resolution optical system (HRME) at baseline, after induction of general anesthesia, and prior to surgery.
  Interventions: Procedure: High-Resolution Microendoscopy; Procedure: Multispectral Imaging; Drug: Proflavine

INTERVENTIONS:
Procedure: High-Resolution Microendoscopy — Undergo evaluation of oral lesions using a high-resolution microendoscope
  Other Names: HRME
Procedure: Multispectral Imaging — Undergo evaluation of oral cavity using a widefield multispectral imaging
Drug: Proflavine — Proflavine) used to stain the mouth tissue after initial imaging.
  Other Names: Proflavine hemisulfate

SUMMARY:
This clinical trial studies wide-field and high resolution in vivo imaging in visualizing lesions in patients with abnormal or uncontrolled oral cell growth (neoplasia) undergoing surgery. Diagnostic procedures, such as wide-field and high resolution in vivo imaging, are devices that let researchers look at a wide area of the lining of the mouth by shining different colors inside the mouth and taking pictures and this may help doctors to decide if a mouth lesion has a high risk of being pre-cancerous or cancerous.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility for assessing oral mucosa in vivo with wide-field and high resolution images obtained using new optical imaging devices composed of cameras and microscopes, and with a topically administered contrast agent.

II. To develop and evaluate algorithms to classify tissue as normal (including hyperkeratosis, hyperplasia, and inflammation) or abnormal (any grade of dysplasia or cancer) based on quantitative parameters extracted from the optical images.

SECONDARY OBJECTIVES:

I. To determine the percentage of subjects and lesions that can be successfully imaged with wide-field and high-resolution optical microscopes after topical application of contrast dye.

II. To identify qualitative and quantitative features within images that differ between pathologically normal, dysplastic, cancerous and inflammatory lesions.

OUTLINE:

Patients undergo evaluation of oral cavity using a widefield multispectral imaging device and a high-resolution optical system (high-resolution microendoscope [HRME]) at baseline, after induction of general anesthesia, and prior to surgery.

After completion of study, patients are followed up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects with oral lesions undergoing surgical resection (i.e., only patients who are scheduled to undergo a surgery of the head & neck area to remove or biopsy oral lesions will be eligible to participate in the study); patients with previous treatment are eligible
* Ability to understand and the willingness to sign a written informed consent document (ICD)

Exclusion Criteria:

* Known allergy to proflavine or acriflavine
* Pregnant or nursing females
* The participant will be excluded from participation in another clinical research trial (i.e., a trial in which an agent is actively administered to the study subject), while being imaged (on active treatment) on this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2010-12-30 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of oral mucosa to be used for non-invasive detection and diagnosis with the use of optical imaging after administration of the topical contrast agent proflavine. | 1 day
  Images obtained will be compared against the histology slides of tissue taken from the same region.
Classification of tissue | 1 day
  Classification algorithms will be developed to separate imaged tissue into 2 diagnostic categories: normal non-neoplastic mucosa vs. dysplasia and cancer

SECONDARY OUTCOMES:
Percentage of subjects and lesions that can be successfully imaged with wide-field and high-resolution optical microscopes after topical application of contrast dye | 1 day
  The data analysis will be descriptive and exploratory in nature. The potential association between sites within the same subject will be examined as well. Performance will be characterized in terms of sensitivity, specificity, area under the ROC curve, and classification accuracy within each diagnostic category.
Qualitative features within images that differ between pathologically normal, dysplastic, cancerous and inflammatory lesions | 1 day
  Performance will be characterized in terms of sensitivity, specificity, area under the ROC curve, and classification accuracy within each diagnostic category.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Gillenwater, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org